CLINICAL TRIAL: NCT02318030
Title: CNTRP Paediatric Outcomes in Transplant: Personalising Immunosuppression to Improve Efficacy (POSITIVE Study)
Brief Title: CNTRP POSITIVE Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Children's Hospital (Other); Stollery Children's Hospital (Other); St. Justine's Hospital (Other); The Children's Hospital of Winnipeg (Other); Montreal Children's Hospital of the MUHC (Other); Provincial Health Services Authority British Columbia (Other); Toronto General Hospital (Other); Vancouver General Hospital (Other); Royal Victoria Hospital, Canada (Other); The Ottawa Hospital (Other); Foothills Medical Centre (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Seema Mital, Staff Cardiologist, The Hospital for Sick Children
Other Study IDs: 1000045186
Record Dates: First submitted 2014-11-25; First posted 2014-12-17 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Transplant; Adaptive Immunity; EBV; Medication Adherence; PTLD
Keywords: Transplant; Adaptive Immunity; EBV; Medication Adherence; Tacrolimus; PTLD
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Immune function testing: blood Pharmacokinetic testing: blood EBV/PTLD viral sequencing: blood EBV/PTLD immunoassays: blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Solid organ transplant
- Hematopoietic Stem Cell Transplant

SUMMARY:
Adequate control of immunosuppression is critical in preventing graft failure after solid organ transplantation (SOT) and in avoiding life-threatening viral and malignant complications. Prolonging patient and graft survival and delaying re-transplantation as children reach adulthood is critical to optimal use of a scarce resource. This requires tailoring post-transplant management to the unique needs of the child. Immunosuppression management is challenging in infants, children and youth. The interval from birth to young adulthood sees profound changes in physiological processes, body size and immune maturation; infancy and adolescence are the periods of most rapid and dramatic change. Three pivotal factors affect immunosuppression control in the child: 1) age-dependent variation in drug metabolism; 2) developmental changes in immune function with increased childhood susceptibility to infections, including those caused by viruses; and 3) behavioural changes in adolescence and young adulthood linked with poor treatment adherence.

This project will identify the most important factors influencing immunosuppression control across the pediatric age range, from infancy to young adulthood, including age-related changes in drug metabolism, immune function, and susceptibility to viral infections, as well as health care system factors affecting treatment adherence. This is the first comprehensive, multi-organ transplant study to identify age-related biologic and health care systems determinants of variability in immunosuppression control in children and youth. Results will inform personalized age-appropriate strategies to improve immunosuppression control and reduce the unacceptably high graft failure and viral complication rates in this vulnerable population.

The POSITIVE Study brings together researchers across Canada and is one of 6 projects and 3 cores that constitute the Canadian Institute of Health Research (CIHR) funded interdisciplinary research program called the Canadian National Transplant Research Program (CNTRP). The CNTRP is a national program designed to increase organ and tissue donation in Canada and enhance the survival and quality of life of Canadians who receive transplants. As a national program, CNTRP provides robust power for pediatric studies that would not otherwise be possible. While primarily focused on issues unique to a pediatric and young adult population, this study will interact closely with all other CNTRP projects. These reciprocal interactions will accelerate new discovery that can be cross-applied in different populations outside of pre-specified age groups. Interactions will ensure rapid knowledge transfer, uptake and dissemination into practice. This is the largest national cohort study of pediatric transplant patients to date in Canada, and it will create a longitudinal dataset with clinical and biological specimens linkable to transplant registries and provincial administrative datasets.

DETAILED DESCRIPTION:
The overall objective of this project is to analyze physiological factors that impact immune response and effect of immunosuppression across different pediatric age groups, to develop age-appropriate medical and health care strategies that can improve graft survival and reduce complications in a pediatric and young adult population. There are 3 primary aims of this study:

Aim 1: Develop age-appropriate calcineurin inhibitor (CNI) dosing for pediatric SOT patients: We hypothesize that physiologically-based (PB) modeling will enable personalized CNI dosing for infants, children and youth based on age, pharmacogenotype and immune maturity. Aim 1 deliverables include 1) a personalized physiologically-based CNI dosing algorithm in SOT; 2) validation of pediatric sensitive immunosuppression monitoring tools and their therapeutic targets; and 3) validation of immunologic assays for assessing age-specific immune responses. We anticipate that personalized CNI dosing will result in early attainment and maintenance of therapeutic drug concentrations, reduce the frequency of out-of-range concentrations post-transplant, improve safety and efficacy of immunosuppression, and reduce dependence on therapeutic drug monitoring to guide drug dosing. Standardized assessment of immune function may also monitor immunosuppression more reliably and eventually reduce the need for invasive monitoring like biopsies.

Aim 2: Develop risk prediction tools based on viral-host interactions that predispose young SOT and hematopoietic stem cell transplant patients to Epstein-Barr virus disorders/post-transplant lymphoproliferative disorder (EBV disorders/PTLD): We hypothesize that susceptibility to EBV disorders/PTLD is influenced by the interaction of high-risk EBV subtypes with host factors like age, immune maturation and intensity of immunosuppression. In the above context, "EBV disorders" refers to non-malignant EBV disease as well as sustained elevation of viral loads in the absence of PTLD. We will identify high-risk viral subtypes and age-related differences in host immunity that interact to increase susceptibility to EBV disorders/PTLD in young patients. Important clinical applications are: 1) knowledge of host susceptibility factors (age and immune maturation) at the time of transplant may assist choice of less intensive immunosuppression to reduce risk of developing EBV (e.g., avoidance of T cell depletion therapies, primary prevention) and promote use of EBV prophylaxis in at risk patients (secondary prevention); 2) an EBV genotype panel will be developed as a clinical tool for detecting high risk subtypes in patients with EBV. This will help identify patients exposed to EBV who should receive aggressive therapy for EBV and/or PTLD (personalized therapy). This innovative risk stratification will enable personalized immunosuppression strategies and strategies to prevent and treat EBV/PTLD.

Aim 3: Develop health care systems strategies to enhance medication adherence in adolescents and young adults: Medication adherence is determined by factors at a variety of different "levels": patient-level (patient-, condition-, and therapy-related factors), "micro"-level (social factors and interactions with the care team), "meso"-level (organization and expertise of the healthcare team and care processes), and "macro"-level (high-level healthcare systems factors, including care and medication cost coverage, and overall care environment). We hypothesize that there are significant differences in modifiable meso- and macro-level systems factors between pediatric programs, between adult programs, and between pediatric and adult programs. Furthermore, we hypothesize that modifiable meso- and macro-level systems factors are independently associated with medication adherence. This aim has two primary objectives:

Objective 1: To characterize differences between Canadian solid organ transplant programs in potentially modifiable meso- and macro-level systems factors.

Objective 2: To identify potentially modifiable meso- and macro-level factors that are determinants of adherence, adjusting for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

Aim 1

* Listed for or recipient of solid organ transplant
* Planned immunosuppression with oral or enteral tacrolimus post-transplant

Aim 2

* Solid organ transplant or hematopoietic stem cell transplant recipients <18 years old
* New onset primary EBV during the first year post transplant (either Donor EBV seropositive, recipient EBV seronegative (D+R-) or donor and recipient seronegative (D-R-) at time of transplant) or new onset EBV/PTLD in the first post-transplant year.
* HSCT patients who develop secondary EBV within the first post transplant year.

Aim 3

* Single organ, kidney, liver, and heart recipients that are at least 3 months post-transplant and 2 months post hospital discharge
* Intact graft function (not currently listed for re-transplant for any organ type or on dialysis
* Receiving maintenance immunosuppression

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: End stage organ failure, Solid organ transplant
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Tacrolimus trough blood concentrations | 1 year from time of transplant
Time to attain stable therapeutic tacrolimus trough blood concentration | 1 year from time of transplant
  Stable therapeutic blood concentration defined as two levels in target therapeutic range without change in dose.
Frequency of out-of-range trough levels during follow-up | 1 year from time of transplant
  Blood concentrations will be captured at 36-48 hours post tacrolimus initiation after transplant, 7, 14, and 30 days after and 3 months and 12 months post transplant.
Determination of trough target therapeutic range | 1 year from time of transplant
  Blood concentrations will be captured at 36-48 hours post tacrolimus initiation after transplant, 7, 14, and 30 days after and 3 months and 12 months post transplant.
Viral genotype | 1 year from time of transplant
  Relationship between major EBV subtypes and clinical and virologic outcomes (illness severity, viral loads, PTLD), evaluated in age groups of <2 years, 2-10 years, 11-18 years and adults >18 years
Taking Adherence to immunosuppressive medications measured using pharmacy refill data and structured self-report | 6 months from a minimum of 3 months post time of transplant
  Participant pharmacies will be contacted at end of study to determine if medications are being refilled as would be expected if all doses were consumed as prescribed.
Immune maturation across pediatric age groups | Baseline & 1 year from time of transplant
Functional immunoassay | 1 year from time of transplant
  Baseline & 1 year from time of transplant
Change in immune function before and after transplant as it correlates with immune maturation and intensity of immunosuppression | Baseline & 1 year from time of transplant
Viral immunoassays | Baseline & 1 year from time of transplant

SECONDARY OUTCOMES:
Graft rejection | 1 year from time of transplant
Complications (cancer, infections, CVS, CNS, other | 1 year from time of transplant
Graft outcomes | Baseline, 3 months, 6 months
Adverse events | Baseline, 3 months, 6 months
Timing adherence to immunosuppressive medications | 6 months from a minimum of 3 months post time of transplant
  Proportion of doses taken late by >25% of the prescribed inter-dose interval
Drug Holidays for immunosuppressive medications | 6 months from a minimum of 3 months post time of transplant
  Period during which 2 or more consecutive doses were missed

CONTACTS AND LOCATIONS:
Overall Officials: Seema Mital, MD, Principal Investigator — SickKids Hospital
Locations (1):
- SickKids Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Papaz T, Allen U, Blydt-Hansen T, Birk PE, Min S, Hamiwka L, Phan V, Schechter T, Wall DA, Urschel S, Foster BJ, Mital S. Pediatric Outcomes in Transplant: PersOnaliSing Immunosuppression To ImproVe Efficacy (POSITIVE Study): The Collaboration and Design of a National Transplant Precision Medicine Program. Transplant Direct. 2018 Nov 27;4(12):e410. doi: 10.1097/TXD.0000000000000842. eCollection 2018 Dec. PMID 30584591
- [Result] Min S, Papaz T, Lambert AN, Allen U, Birk P, Blydt-Hansen T, Foster BJ, Grasemann H, Hamiwka L, Litalien C, Ng V, Berka N, Campbell P, Daniel C, Saw CL, Tinckam K, Urschel S, Van Driest SL, Parekh R, Mital S. An Integrated Clinical and Genetic Prediction Model for Tacrolimus Levels in Pediatric Solid Organ Transplant Recipients. Transplantation. 2022 Mar 1;106(3):597-606. doi: 10.1097/TP.0000000000003700. PMID 33755393
- [Result] Dabirzadeh A, Dahhou M, Zhang X, Sapir-Pichhadze R, Cardinal H, White M, Johnston O, Blydt-Hansen TD, Tibbles LA, Hamiwka L, Urschel S, Birk P, Bissonnette J, Matsuda-Abedini M, Harrison J, Schiff J, Phan V, De Geest S, Allen U, Mital S, Foster BJ. Care processes and structures associated with higher medication adherence in adolescent and young adult transplant recipients. Pediatr Transplant. 2021 Dec;25(8):e14106. doi: 10.1111/petr.14106. Epub 2021 Aug 2. PMID 34339090